CLINICAL TRIAL: NCT07353996
Title: Determination of the Effective Dose of a Single Intravenous Dose of Tegileridine Fumarate for Postoperative Analgesia After Orthopedic Surgery: A Up-and-Down Sequential Allocation Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0393
Record Dates: First submitted 2025-12-24; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single intravenous Tegileridine Fumarate arm (Experimental)
  Interventions: Drug: Single intravenous injection of Tegileridine Fumarate

INTERVENTIONS:
Drug: Single intravenous injection of Tegileridine Fumarate — Single intravenous injection of tegileridine fumarate for postoperative analgesia in adult patients (18-75 years, ASA I-III) undergoing orthopedic surgery, including spinal fusion, femoral fracture fixation, and total knee arthroplasty. The study uses a dose-escalation design to determine the 90% effective dose (ED90).
  Doses: To be determined using an up-and-down sequential allocation method (dose-ranging study).

SUMMARY:
The goal of this clinical trial is to determine the 90% effective dose (ED90) of a single intravenous injection of tegileridine fumarate for postoperative analgesia in adult patients aged 18-75 years with American Society of Anesthesiologists (ASA) physical status I-III undergoing orthopedic surgery, including spinal fusion surgery, femoral fracture fixation, and total knee arthroplasty.

The main questions this study aims to answer are:

What is the ED90 of a single intravenous dose of tegileridine fumarate for achieving adequate postoperative analgesia, defined as a Numeric Rating Scale (NRS) pain score ≤ 3 within 30 minutes after awakening from anesthesia without the need for rescue analgesia?

Participants will:

Receive a single intravenous injection of tegileridine fumarate during skin closure at the end of surgery.

Start with an initial dose of 0.5 mg, with subsequent doses adjusted upward or downward in 0.1 mg increments for the next participant based on the analgesic response of the preceding participant, following a biased-coin up-and-down sequential dose allocation design.

Be closely monitored during the postoperative recovery period for pain intensity, vital signs (including heart rate, blood pressure, respiratory rate, and oxygen saturation), and adverse reactions such as nausea, vomiting, respiratory depression, agitation, and other opioid-related side effects.

This study aims to identify an optimal single-dose regimen of tegileridine fumarate that provides effective postoperative analgesia with an acceptable safety profile, thereby improving postoperative pain control and promoting enhanced recovery in patients undergoing orthopedic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 75 years.
* Scheduled for elective orthopedic surgery, including spinal fusion, femoral fracture fixation, or total knee arthroplasty.
* American Society of Anesthesiologists (ASA) physical status I-III.
* Ability to understand the study procedures and provide written informed consent.

Exclusion Criteria:

* Patients with moderate to severe obesity (BMI > 30 kg/m²).
* Known hypersensitivity or allergy to tegileridine fumarate or other analgesics.
* History of chronic pain or long-term use of opioids.
* Severe hepatic or renal impairment.
* Patients requiring postoperative ICU care.
* Severe respiratory depression (e.g., oxygen saturation < 90%).
* Known or suspected gastrointestinal obstruction, including paralytic ileus.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-10-25 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Effective dose producing adequate postoperative analgesia in 90% of patients (ED90) | Within 30 minutes after awakening from anesthesia
  The primary outcome was the 90% effective dose (ED90) of a single intravenous bolus of tegileridine for postoperative analgesia following orthopedic surgery. Analgesic success was defined as a Numeric Rating Scale (NRS) pain score ≤ 3 within 30 minutes after awakening from anesthesia without the need for rescue analgesics.
  Dose allocation followed a biased-coin up-and-down sequential design, with dose adjustments based on the analgesic response of the preceding patient. The ED90 and its 90% confidence interval were estimated using isotonic regression analysis.

SECONDARY OUTCOMES:
Incidence and severity of postoperative nausea and vomiting (PONV) | From drug administration to 24 hours postoperatively
  The incidence and severity of postoperative nausea and vomiting (PONV) within 24 hours after administration of tegileridine were assessed. PONV was evaluated by trained clinical staff using a standardized ordinal severity scale, defined as:
  0 = no nausea or vomiting;
  1. = nausea only;
  2. = retching (dry heaves);
  3. = vomiting.
Heart rate (HR) | From immediately before drug administration to 24 hours postoperatively
  Measured in beats per minute (bpm).
Respiratory Rate (RR) | From immediately before drug administration to 24 hours postoperatively
  Measured in breaths per minute (bpm).
Peripheral Oxygen Saturation (SpO₂) | From immediately before drug administration to 24 hours postoperatively
  Measured as a percentage (%).
Extubation-related airway responses | From extubation until 10 minutes after extubation
  Incidence of airway reactions during emergence from anesthesia, including coughing and laryngospasm, assessed by the attending anesthesiologist at the time of tracheal extubation.
Postoperative rescue analgesia requirement | From awakening to 24 hours postoperatively
  Use of rescue analgesia after surgery, including whether additional opioid analgesics were required within 30 minutes after awakening and cumulative opioid consumption within 24 hours postoperatively (converted to morphine equivalents).
Patient-controlled analgesia (PCA) usage | From awakening to 24 hours postoperatively
  PCA usage parameters, including number of effective and total PCA button presses and total PCA-delivered opioid dose within 24 hours after surgery.
Postoperative pain intensity (NRS scores) | 30 minutes, 6 hours, 12 hours, and 24 hours after awakening
  Pain intensity assessed using the Numeric Rating Scale (NRS, 0-10; 0 = no pain, 10 = worst imaginable pain) at rest and during movement at predefined postoperative time points.
Incidence of postoperative adverse events | From drug administration to 24 hours postoperatively
  Incidence of adverse events, including agitation (Richmond Agitation-Sedation Scale ≥2), delirium (Nu-DESC score ≥2), respiratory depression (SpO₂ <90%), delayed emergence, pruritus, dizziness, shivering, and postoperative nausea and vomiting (PONV), graded according to severity.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University anesthesiology department, Hanzhong, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No